CLINICAL TRIAL: NCT04070040
Title: An Exploratory Study on Camrelizumab（SHR-1210）for Recurrent Primary Central Nervous System Lymphoma (PCNSL)
Brief Title: Camrelizumab for Patients with Recurrent Primary Central Nervous System Lymphoma (PCNSL)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Sanbo Brain Hospital (Other)
Responsible Party: Principal Investigator, Junping Zhang, Beijing Sanbo Brain Hospital, Beijing Sanbo Brain Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1.0
Record Dates: First submitted 2019-08-25; First posted 2019-08-28 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Primary Central Nervous System Lymphoma
MeSH Terms: interventions — camrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Camrelizumab (Experimental): Camrelizumab(SHR-1210) 200mg, once every 2 weeks, each 4 weeks is 1cycle.
  Interventions: Drug: Camrelizumab

INTERVENTIONS:
Drug: Camrelizumab — Camrelizumab(SHR-1210) 200mg, once every 2 weeks, each 4 weeks is 1cycle.
  Other Names: SHR-1210

SUMMARY:
This study is intend to improve the objective response rate in treatment of camrelizumab in recurrent primary central nervous system lymphoma patients.

DETAILED DESCRIPTION:
Primary CNS lymphoma (PCNSL) is a rare B-cell variant of non-Hodgkin lymphoma that is confined to the brain, leptomeninges, spinal cord, and eyes. The optimum treatment for patients with recurrent PCNSL remains challenging and at present there is no universally accepted therapeutic approach . The purpose of this study is to evaluate the efficacy and safety of camrelizumab [a programmed cell death 1 (PD-1) inhibitor] for recurrent patients with primary CNS lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. The initial diagnosis was primary diffuse large B-cell lymphoma of the central nervous system confirmed by histopathology;
2. Prior to first-line treatment based on methotrexate (with or without radiotherapy), tumor recurrence was confirmed by MRI;
3. Measurable focus in MRI (>10x10mm);
4. Aged > 18 years;
5. Life expectancy of at least 12 weeks;
6. The patient has a Karnofsky performance status of at least 50%;
7. Main organs function normally, without serious blood, heart, lung, liver, kidney and immune deficiency diseases. Specific assay indicators requirements： White blood cells>3.0×10^9/L;platelet>80×10^9/L;hemoglobin>10g/dL;serum bilirubin ≤ 1.5×ULN;ALT and AST ≤ 2×ULN;serum creatinine≤1.5mg/dL;
8. Female subjects of childbearing age must exclude pregnancy and are willing to use a medically approved high-efficiency contraceptive (eg, IUD, contraceptive or condom) during the study period and within 3 months of the last study drug administration;
9. The subject should be aware of the purpose of the study and the operations required by the study and volunteer to participate in the study before sign the informed consent form;

Exclusion Criteria:

1. Concurrent administration of any other antitumor therapy；
2. Allergic to the ingredients of research drugs；
3. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent；
4. Any active autoimmune diseases or a history of autoimmune diseases (including but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, nephritis, hyperthyroidism, decreased thyroid function；
5. Systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment, except for a maximum dose of 4 mg/day dexamethasone or equivalent doses of other corticosteroids or control of brain edema, which has been stable or decreased for at least 1 week prior to inclusion;
6. Active infection;
7. Risk of bleeding;
8. HIV positivity;
9. Pregnancy and lactation;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2020-02-13 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR(objective response rate) | Up to three years
  the proportion of patients with tumor size reduction of a predefined amount and for a minimum time period

SECONDARY OUTCOMES:
The best therapeutic response of CR(complete response)、PR(partial response)、SD(stable response) and PD(progressive disease) | Up to three years
  Describe the best therapeutic response of patients treated with Camrelizumab
PFS(progression free survival) | Up to three years
  the time from randomization until objective tumor progression or death
OS(overall survival) | Up to three years
  the time from randomization until death from any cause and is measured in the intent-to-treat population
ADEs( adverse events) | Up to three years
  Adverse events at each visit with the NCI CTCAE v5.0 used as a guide for the grading of severity.
KPS(Karnofsky Performance Status) | Up to three years
  Duration of stabilization/improvement of Karnofsky Performance Status

CONTACTS AND LOCATIONS:
Locations (1):
- Sanbo Brain Hospital Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No